CLINICAL TRIAL: NCT00202592
Title: Safety and Effects on Blood Pressure of Daily Dose 0.025 to 0.135 Milligram Per Kilogram of S90625 a Paediatric Formulation of Perindopril, in Hypertensive Children - 24 Months
Brief Title: S90652 in Paediatric Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut de Recherches Internationales Servier (Other)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: CL2-90652-002
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Perindopril

INTERVENTIONS:
Drug: Perindopril

SUMMARY:
The aim of the study is to assess the long-term safety and effects on blood pressure of a paediatric formulation of perindopril in hypertensive children

ELIGIBILITY:
Inclusion Criteria:

* Hypertensive children, who have been treated for four months at least with S90652, with safety and efficacy

Exclusion Criteria:

* Poorly controlled hypertension
* Girls with signs of pubescence

Ages: 30 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2003-11; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Clinical safety assessed from the patient's (parents) complaints and clinical follow-up

SECONDARY OUTCOMES:
Blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Niaudet, Pr, Study Chair — Hôpital Necker-Enfants Malades, Paris, France
Locations (1):
- Hôpital Necker Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Researchers can ask for a study protocol, patient-level and/or study-level clinical trial data including clinical study reports (CSRs).
  They can ask all interventional clinical studies in patients:
  * submitted for new medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * Where Servier or an affiliate are the Marketing Authorization Holders (MAH). The date of the first Marketing Authorization of the new medicine (or the new indication) in one of the EEA Member States will be considered within this scope.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorisation in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: http://clinicaltrials.servier.com